CLINICAL TRIAL: NCT07111858
Title: Pavlik Harness Treatment Versus Monitoring for Treatment of Graf Type 2b and 2c Hip Developmental Dysplasia of the Hip (DDH)
Brief Title: Pavlik Harness Treatment vs Monitoring for Treatment of Developmental Dysplasia of the Hip (DDH) in Babies Diagnosed With Graf Type 2 Hips
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Principal Investigator, Nicole Hilburn, Senior Lecturer, Canterbury Christ Church University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 304944
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Developmental Hip Dysplasia
Keywords: DDH
MeSH Terms: conditions — Developmental Dysplasia of the Hip | interventions — Watchful Waiting; Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pavlik Harness Treatment (No Intervention): This is usual care with a Pavlik Harness
- Watchful waiting and regular ultrasound scans (Experimental): Watchful waiting, with ultrasound scans every 3 weeks
  Interventions: Other: Watchful waiting with supportive care

INTERVENTIONS:
Other: Watchful waiting with supportive care — Usual care is Pavlik Harness Treatment. Watchful waiting with ongoing ultrasound scans is the intervention in this study to determine whether the hip matures without the use of the Pavlik Harness
  Arms: Watchful waiting and regular ultrasound scans

SUMMARY:
Developmental Dysplasia of the Hip (DDH) is thoroughly manageable if treated correctly. While the standard treatment is using a Pavlik harness, there is not enough research regarding those patients who have stable but immature Graf type 2b and 2c hips and whether a harness is needed.

At Maidstone and Tunbridge Wells NHS Trust, all babies who present with Graf type 2b and 2c hip dysplasia are treated using a Pavlik harness, which is worn 24 hours a day for up to 12 weeks. Although the harness is usually very comfortable, it can result in stress and anxiety for parents, and may make caregiving activities such as bathing, feeding and carrying more difficult.

Our aim is to run a feasibility trial, recruiting babies with type 2b and 2c hip dysplasia, to determine whether there is any difference in a group which is treated with Pavlik harnessing, or whether these hips do in fact mature on their own. We would like to ensure that Pavlik harness treatment is indeed necessary in these groups.

Babies randomised to the comparator group with type 2b and 2c hips would be treated using a Pavlik Harness and following the usual protocol with ultrasound scans at 3 weeks, 8 weeks and 12 weeks post start of treatment, and harness duration is determined by the scan at 8 weeks.

Babies randomised to the Intervention group would be monitored via ultrasound scans at 3 weeks, 6 weeks, 8 weeks and 12 weeks post diagnosis, and should it be determined that their hips are not maturing spontaneously, they will be placed in a harness immediately, and follow the treatment-group protocol. Since the scans are done so frequently, and their hips are stable, there is no risk to these babies.

Babies in both groups would have x-rays at 9 months and 15 months to determine longer-term outcome.

The trial will last for 15 months after diagnosis for each patient, and the end-point of the study would be on achieving a 15-month x-ray for the last recruited patient.

Patients will be informed of the results of the study.

DETAILED DESCRIPTION:
Developmental dysplasia of the hip (DDH) is a common cause of childhood disability, and diagnosis after 3 months may lead to the need for surgery and long-term complications. The incidence in the UK before ultrasound (US) screening became available was 1-2 per 1000. Since the advent of selective US screening, estimates in the UK incidence range from 5-30 per 1000. In terms of criteria for screening, there is consensus that a family history of DDH, female gender, breech presentation, primiparity and oligohydramnios increase the risk of DDH, although screening criteria vary amongst centres. There is a lack of evidence to support birth weight, prematurity, multiple pregnancy, mode of delivery or the presence of foot deformity as increased risk-factors for DDH.

Radiographic depiction of the hip is difficult in the first few months of life, due to the absence of the ossific nucleus. The advent of ultrasound (US) has significantly impacted these challenges, and this method has become popular since the first paper describing it by Graf in 1980. The Graf method has been accepted as the Gold Standard in Ultrasound analysis.

Differences in image acquisition and interobserver variation can significantly influence the diagnosis in the border zones between the different categories of the classifications. Reviews conclude that diagnosis by US is 'highly sensitive but poorly specific', and it is not clear how much unnecessary treatment is instituted due to the lack of a benchmark for diagnosis. It is unclear in well centered, stable hip dysplasia, whether treatment alters the natural history of the development of the hip. Randomised trials of abduction treatment of dysplastic hips according to the existing classification systems have failed to show a difference between the treatment and non-treatment groups between six weeks and three months, and between three months and six months .

While low risk, the Pavlik harness is not entirely benign. The rate of avascular necrosis (AVN) varies widely according to application , and has been associated with a longer duration of treatment.

While other complications from a correctly applied harness are rare, it may cause skin crease dermatitis and femoral nerve palsy (which has been linked with treatment failure). It is therefore beneficial to keep time spent in a harness to a minimum, and initiate treatment only when necessary.

In a very recent consensus study in which 35% of respondents stated that they treat a stable dysplastic hip in an infant of less than six weeks of age with a flexion/abduction orthosis. Fifty three percent had a treatment threshold (the mildest form of hip pathology deemed to require treatment) of dysplasia at above six weeks of age, and for 11%, the threshold was an unstable or dislocatable hip. There was near universal agreement that subluxed or dislocated but reducible hips require treatment at any age. Forty three percent would attempt to treat a dislocated but irreducible hip with a harness. There were no identifiable trends among those who treat dysplasia under six weeks of age.

Why is this important? Consensus amongst surgeons is crucial to achieve, particularly as parents and carers become more informed through social media, support groups and increased access to information. National programmes such as the United Kingdom's 'Getting It Right First Time' promotes standardisation of care by healthcare providers , and the committee of the Newborn and Infant Physical Examination Programme (NIPE) has indicated that standardisation of diagnosis and treatment pathways would be a prerequisite for establishing a national universal ultrasound screening programme in the United Kingdom. The Steps charity has called for consensus in order to manage parental angst in discussion forums, as variation in screening and treatment protocols may lead to increased anxiety. The NIPE committee has suggested that standardisation of treatment may be the basis on which to better integrate hip dysplasia into national screening pathways.

There is unnecessary variation in the treatment of infantile DDH. This variation is preventing the United Kingdom national screening programme adopting standards for reporting within their NIPE-Smart system as the correct treatment pathway is uncertain. Furthermore, the uncertainty may contribute to the apparent failure of screening within the UK compared to other healthcare systems. Due to the fact that treatment consensus is lacking particularly in the group with well-centred, stable dysplastic hips, this study aims to investigate Pavlik harness treatment versus active surveillance in acetabular development in these babies. If successful, this research will lead to an adequately powered randomised control trial to inform policy, contribute to the development of treatment consensus, and provide evidence for best practice for this group of patients.

A total of 70 subjects will be recruited across the Maidstone and Tunbridge Wells sites. This will be in collaboration with the ultrasonographers who conduct screening ultrasounds weekly with clinic support as necessary

6.1 Reliability

Reliability in measuring ultrasound will be run between the ultrasonographers and consultants whose clinics the babies will be recruited from on 5 babies per pair. A kappa coefficient of 0.9 to 1 would be deemed acceptable.

Reliability of harness fitting and checks would be run between the consultant and the member of staff responsible for fitting the harnesses to ensure a standard fitting and harness check protocol.

6.2 Screening and eligibility assessment

Potentially eligible participants will be identified by the ultrasonographers following screening ultrasounds, and a Graf classification of 2b or 2c. The baby will be booked into a consultant clinic, and the ultrasound results will be confirmed by the consultant. Screening logs will be kept at each site to determine the number of patients assessed for eligibility and reasons for exclusion. In addition, the number of eligible and recruited patients, and the number of patients who decline consent or withdraw will be recorded.

6.3 Informed consent

A member of the responsible clinical team will briefly highlight the study to the patient's parent. They will approach the patient, or contact them via telephone if they are unable to meet the patient face-to-face, and explain the trial. In order to standardise the information provided to the patients, online and written recruitment materials will be made available to the parent This will then lead on to an informed consent discussion, which would place take in person. Patients will be given as much time as possible to consider the information and discuss it with relatives/carers. It will be clearly stated that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, without affecting their legal rights, and with no obligation to give the reason for withdrawal.

Prior to any study-related procedures or data being collected participants parent/carer will complete the latest approved version of the consent form and provide their contact details if they are willing to consent in order for an electronic copy of the form to be sent to them immediately. The person who obtained the consent must be suitably qualified and experienced and have been authorised to do so by the Principal Investigator. Once completed, an electronic version of the signed consent form will be automatically emailed to the participant. The local research team will be able to download a copy to place in the participant's medical notes. If the participant does not have access to email then a paper copy of their consent form will be provided by the local research team instead.

6.4 Randomisation

Once informed consent has been given, the patient will be randomised to the surveillance or harness group using a validated computer randomisation program.

6.5 Description of study procedures

Participants will be randomised to receive either Pavlik harness treatment or active surveillance. This will be under the supervision of a consultant trauma and orthopaedic surgeon.

6.6 Baseline assessment

The initial ultrasound scan will form the basis for the baseline assessment, and a thorough history and clinical examination will be performed. This will include a hip examination, general examination to exclude other medical issues such as a sacral dimple, torticollis and any evidence of neurological problems. This will all be documented in the patient notes, and transferred to a database. The parenting stress index form would be administered at baseline to both groups.

6.7 Harness application

A Pavlik harness will be applied to the babies in the treatment group by (specify person), and all information around harness care and treatment given to the parent/caregiver. A contact number is provided should any concerns around the harness arise. The baby's harness is checked at 1 week, 3 weeks, 6 weeks and 9 weeks post diagnosis to ensure that it is fitting correctly, and a new size is not needed. This is done by the consultant or one of 3 orthopaedic Extended Scope Practitioner (ESP) physiotherapists. Skin condition, femoral nerve integrity and flexion/abduction position of the hips are checked at these points. At week 3 the PSI-SF is administered which will help to determine stress levels of the parent/caregiver and provide appropriate support as required. Ultrasound scans are performed at 3, 6, 9 and 12 weeks, and will be measured and interpreted by both the ultrasonographer and the consultant. The parent is given an emergency contact number for the team at the initial appointment, for any issues with the harness. This contact number provides the parent with access to support from the DDH team for any issues they may encounter, as well as any support the parent/guardian needs. There are 3 hip clinics per week which they are able to drop into, and if they need to be seen urgently, an appointment would be made specifically for this (standard care). Should the ultrasound results not demonstrate Graf 1 mature hips bilaterally by 12 weeks in a Pavlik harness, the baby is placed in an abduction splint for night and nap time, until their x ray at 9 months of age (standard care).

6.8 Surveillance group

This group receives no harness, but will be scanned using ultrasound at 3 weeks, 6 weeks, 9 weeks and 12 weeks, and measured and interpreted by both the ultrasonographer and consultant. The PSI-SF will be administered at 3 weeks which will help to determine stress levels of the parent/caregiver so this can be compared with the harness group. Should the ultrasound scan at 3 weeks not show any maturation of the hip/s, the baby would be placed in a harness and into the treatment group with appropriate documentation for analysis. The same emergency number is given to parents in this group for any concerns that may arise between appointments, as well as to provide any support that the parent/guardian needs.

6.9 Parent/caregiver focus groups Two parent/caregiver focus groups will be run during the course of data collection to obtain qualitative data around experiences of having a baby who has a diagnosis of DDH, the information and support received during the treatment period, as well as experiences of being in either the harness group or the monitoring group. One group will consist of parents/caregivers whose babies were in the non-harness group and the second focus group will consist of parents/caregivers whose babies were in the harness group. These groups will be conducted on Microsoft Teams, lasting approximately 1.5 to 2 hours, and will be recorded. Data will be analysed using NVivo.

Parents whose babies have completed the treatment period will be eligible to attend, and will be given an information sheet, and invited to have any questions answered before completing a consent form, and being included in the group. Parents will be able to withdraw prior to the start of the focus group, but will be informed that data cannot be removed from the discussion on completion of the group (this is outlined within the information sheet as well). A discussion guide is attached as an appendix to the protocol.

ELIGIBILITY:
Inclusion Criteria:

•Infants from birth to 16 weeks with Graf type 2b or 2c hip dysplasia on ultrasound

Exclusion Criteria:

* associated neuromuscular, genetic or neurological condition which may complicate the course of treatment
* babies who have unstable hips on clinical examination

Ages: 0 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Ultrasound | 12 weeks after baseline scan
  An alpha angle of 60 degrees using Graf Classification needs to be obtained to denote a normal hip
Ultrasound | 12 weeks after initial scan
  Alpha angle of 60 degrees needs to be obtained using the Graf classification in order to denote a normal hip

SECONDARY OUTCOMES:
Parenting Stress Index | 3 weeks after baseline scan
  Questionnaire to determine stress levels of parents whose babies are in the harness and non-harness groups
X Ray | 9 months and 15 months of age
  X ray to determine Acetabular Index at 9 months and and 15 months of age to determine whether the hip is normal once the baby starts weightbearing

CONTACTS AND LOCATIONS:
Locations (1):
- Maidstone and Tunbridge Wells NHS trust, Royal Tunbridge Wells, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollet V, Sakkers R, Beek E, et al. Abduction bracing versus natural history in hip dysplasia: multicenter randomized trial. J Child Orthop 2016;10:S30-S31
- [Background] Bracken J, Ditchfield M. Ultrasonography in developmental dysplasia of the hip: what have we learned? Pediatr Radiol. 2012 Dec;42(12):1418-31. doi: 10.1007/s00247-012-2429-8. Epub 2012 Sep 2. PMID 22940710
- [Background] Abidin, R. R. (1995). Parenting Stress Index. Lutz, Florida: Psychological Assessment Resources, Inc.